CLINICAL TRIAL: NCT05726669
Title: Randomised Controlled Trial of Self-help Cognitive Behavioural Therapy for Depression in Adults With Pulmonary Hypertension.
Brief Title: Self-help Booklets for Depression in Adults With Pulmonary Hypertension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Abbie Stark, Principal Investigator, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHDEP2023
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Hypertension; Depression
MeSH Terms: conditions — Hypertension, Pulmonary; Depression

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial (RCT) design will be used, with participants randomised on a 1:1 basis to either a CBT informed self-help intervention to help manage depression in pulmonary hypertension or a controlled wait list condition.
Masking Description: Both participants and researchers will not be blinded to condition. This is necessary as participants will know before they consent to the study that they may be randomised to a wait list condition or the intervention, and the lead researcher will contact participants during the intervention (at two weeks) to gather acceptability and adherence feedback. Therefore the researcher needs to know who is in the intervention group to contact them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Self-help intervention based on cognitive behavioural therapy for depression in pulmonary hypertension. There will be four booklets which will take four weeks for participants to work through in their own time at home.
  Interventions: Other: Self-help materials for depression
- Wait list control group (No Intervention): The wait list control group will not receive the self-help intervention, and will be compared to the intervention group on the outcome measures. The wait-list control group will receive the intervention after study completion if it is found to be helpful (June 2024).

INTERVENTIONS:
Other: Self-help materials for depression — Self-help materials for depression based on cognitive behavioural therapy have been created and tailored to those with PH by researchers involved in this project, using the evidence base and theory plus clinical experience. The Medical Research Council Frameworks for complex interventions (Craig et al., 2008; Skivington et al., 2021) have been followed as well as the quality appraisal tool for self-help interventions in depression (Cape, 2015). The self-help materials will be shared for feedback with a readership panel of people with PH and caregivers who are members of Pulmonary Hypertension Association UK (a charity for people with PH) prior to being given to participants. The self-help materials will be provided online or posted in paper form to the intervention group and will take four weeks for the person to complete at home (one booklet per week).
  Arms: Intervention group

SUMMARY:
The investigators have developed self-help booklets specifically for adults with PH who are experiencing difficulties with depression. The self-help booklets are based on a type of psychological treatment called Cognitive Behavioural Therapy or CBT for short.

* CBT looks at the way people think and what they do, and how this affects their mood.
* It involves making changes to thoughts and behaviours.
* CBT can help people develop more helpful ways of coping with depression.
* CBT is one of the most effective therapies for depression, this means it works well.

There are four booklets that participants will work though weekly in their own time and at home. The aim of this study is to test whether the self-help booklets are helpful in reducing depression in people with pulmonary hypertension.

Those taking part will be asked to complete a series of questions asking about themselves including whether they are experiencing any difficulties such as depression and anxiety.

They will then be allocated at random to one of two groups. Group one will receive the self-help booklets, called the intervention group. Group two, or the wait list group, will receive the intervention at a later date if it is found to be helpful. Having two groups is very important as it will allow us to see whether benefits associated with taking part in the project was because of the self-help booklets or something else.

Participants in group one will also be contacted partway through the intervention to ask about their experiences of taking part.

Both groups will be asked to complete a series of questionnaires four weeks later and then again in one month. Participants in group one will be contacted again to find out more about their experiences of the project.

DETAILED DESCRIPTION:
Previous research has demonstrated high rates of depression in people with pulmonary hypertension (PH). The psychological interventions that support people with depression are not made specific to people with PH and may not be relevant for them, and there is limited evidence examining psychological treatments for depression in people with PH. The aim of this study is to develop and test a self-help psychological intervention for depression based on cognitive behavioural therapy (CBT), which has been developed specifically for individuals with PH. When participants have agreed to take part, they will be allocated at random into an intervention or wait-list group. The self-help materials will be provided online (for people outside of the UK) or posted in paper form (for those living in the UK) and will take four weeks to complete at home. Both groups will complete questionnaires at the same time points (before starting the study, after four weeks and after eight weeks (pre-, post-intervention and one-month follow up). In addition, the intervention group will be contacted after two weeks of their participation and asked about their experiences of the intervention and participation in the study - measuring acceptability of the intervention. The intervention group will also be asked to complete a feedback questionnaire after completing the intervention to further examine acceptability. Analysis will be conducted by the researcher to examine whether the self-help intervention reduced depression in individuals with PH, compared to those with PH who did not receive the intervention. The potential benefit of the study includes a new intervention for depression in people with PH. When the study is completed, if the intervention is found to be helpful and safe, then the people who took part in the study and did not receive the intervention will be offered the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary hypertension
* Over the age of 18 years
* Able to complete questionnaires without help from others
* Can understand English
* They will read all study documents in detail and ask the researcher any questions they have. Based on this, they could provide informed consent to take part if they are eligible.
* Feels like they have difficulties with depression, low mood or negative thoughts.
* Not currently experiencing thoughts of self-harm or suicide. This means that they have not had thoughts of self-harm or suicide within the last month.

Exclusion criteria:

* Current thoughts of self-harm or suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Depression | Pre-, post intervention and one month follow up. This means before starting the study, after 4 weeks and after 8 weeks. Analysis will test if there is a change at baseline, post intervention and follow up between groups.
  The Patient Health Questionnaire (PHQ-8) (Kroenke et al., 2009) will be used to measure depression as the primary outcome. The minimum score is 0 and the maximum score is 24. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Anxiety | Pre-, post intervention and one month follow up. This means before starting the study, after 4 weeks and after 8 weeks. Analysis will test if there is a change at baseline, post intervention and follow up between groups.
  The Generalised Anxiety Disorder (GAD-7) (Spitzer et al., 2006) will be used to measure anxiety. The minimum score is 0 and the maximum score is 21. A higher score indicates a worse outcome.
Health-related quality of life | Pre-, post intervention and one month follow up. This means before starting the study, after 4 weeks and after 8 weeks. Analysis will test if there is a change at baseline, post intervention and follow up between groups.
  The emPHasis-10 (Yorke et al., 2014) will be used to measure health-related quality of life. The minimum score is 0 and maximum score is 50. A higher score indicates a worse outcome.
Fatigue | Pre-, post intervention and one month follow up. This means before starting the study, after 4 weeks and after 8 weeks. Analysis will test if there is a change at baseline, post intervention and follow up between groups.
  The Fatigue Severity Scale (FSS) (Learmouth et al., 2013) will be used to measure fatigue. The minimum score is 9 and the maximum score is 63. A higher score indicates a worse outcome.
Pain Self Efficacy | Pre-, post intervention and one month follow up. This means before starting the study, after four weeks and after eight weeks. Analysis will test if there is a change at baseline, post intervention and follow up between groups.
  The Pain Self-Efficacy Questionnaire (Nicholas, 2007) will measure pain. The minimum score is 0 and the maximum score is 60. A higher score indicates a better outcome.
Cognition and behaviours | Pre-, post intervention and one month follow up.This means before starting the study, after 4 weeks and after 8 weeks. Analysis will test if there is a change at baseline, post intervention and follow up between groups.
  To examine whether cognitions and behaviours have an impact on change in depression, the Cognitive Behavioural Processes Questionnaire (CBP-Q) will be used. The minimum score is 0 and the maximum score is 120. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Stark, Psychology, Principal Investigator — Cardiff University
Locations (1):
- Cardiff University - however recruitment is done electronically, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study investigators aim to publish the final report in a peer reviewed international journal and also make the anonymised data available in Cardiff University's data repository. The investigators would also like to share the findings in conferences. The data in anonymised format would be available to other researchers upon reasonable request. When the study is complete, electronic files will be stored for a minimum of 15 years by Cardiff University after the end of the project or after publication of any findings based upon the data (whichever is later). The end of project is defined as completion of project closure report or publishing of final articles. This follows Cardiff University's research records retention policy.
Supporting Information: Study Protocol, SAP
Time Frame: When the study is complete, electronic files will be stored for a minimum of 15 years by Cardiff University after the end of the project or after publication of any findings based upon the data (whichever is later). The end of project is defined as completion of project closure report or publishing of final articles. This follows Cardiff University's research records retention policy. Data can be made available following study completion, up until the point of disposal of data after 15 years.
Access Criteria: Data will be made available to researchers upon reasonable request.

REFERENCES:
- [Result] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Yorke J, Corris P, Gaine S, Gibbs JS, Kiely DG, Harries C, Pollock V, Armstrong I. emPHasis-10: development of a health-related quality of life measure in pulmonary hypertension. Eur Respir J. 2014 Apr;43(4):1106-13. doi: 10.1183/09031936.00127113. Epub 2013 Nov 14. PMID 24232702
- [Result] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Result] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Result] Learmonth YC, Dlugonski D, Pilutti LA, Sandroff BM, Klaren R, Motl RW. Psychometric properties of the Fatigue Severity Scale and the Modified Fatigue Impact Scale. J Neurol Sci. 2013 Aug 15;331(1-2):102-7. doi: 10.1016/j.jns.2013.05.023. Epub 2013 Jun 20. PMID 23791482
- [Result] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488